CLINICAL TRIAL: NCT07248085
Title: The Effect of Rapid Relaxation Exercise and Cold Application on Pain, Anxiety, and Satisfaction Before Chest Tube Removal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Tülay KILINÇ, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: tulay39
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Open Heart Surgery
Keywords: Chest Tube; Rapid Relaxation Exercise; Cold Application; Pain; Anxiety; Patient Satisfaction
MeSH Terms: conditions — Pain; Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cold Application (Experimental): Cold Application
  Interventions: Other: Cold Application
- Rapid Relaxation Exercise (Experimental): Rapid Relaxation Exercise
  Interventions: Other: Rapid Relaxation Exercise
- Standard care (No Intervention): In our study, no intervention other than the clinical protocol will be applied to the control group patients before chest tube removal.

INTERVENTIONS:
Other: Cold Application — Patients will receive routine monitoring, pharmacological treatment, and nursing care in the unit where the study is conducted. Cold application ice packs will be placed around the patient's chest tube insertion site. The ice pack, which has been kept in the research clinic's refrigerator for 72 hours, measured with a barbeque thermometer at -10°C, and distributed evenly when cooled, will be placed on the chest tube dressing. Since skin temperature must fall below 13.6°C for cold application to have a local analgesic effect, the patient's skin temperature will be measured at one-minute intervals throughout the cold application. When the application reaches 13.6°C, the application will be stopped, and the physician will be notified that the patient is ready. During the cold application, the applied area will be checked for redness, irritation, and discoloration.
  Arms: Cold Application
Other: Rapid Relaxation Exercise — Individuals in the rapid relaxation exercise group will be led by the researcher in the patient room or examination room to perform a breathing exercise. The exercise will last approximately 5-10 minutes. The environment will be quiet, at room temperature, and well-ventilated. The exercises will be performed by ensuring the patient is seated in a comfortable position, and the following steps will be followed. Patients will be asked to close their eyes and observe the up-and-down movement of their abdominal muscles as they breathe in and out. The same exercise will be repeated for seven cycles. Patients are asked to inhale deeply and slowly to revitalize their entire body and feel a sense of lightness. On the exhale, they are asked to completely relax all their muscles by making the sound "A" (A-Kara). Once completely relaxed, they are encouraged to blink their eyes open several times.
  Arms: Rapid Relaxation Exercise

SUMMARY:
A chest tube is inserted to drain air, fluid, or blood from the pleural space and is vital for restoring respiratory function in the postoperative period. However, tube removal is often described by patients as one of the most painful and anxiety-provoking experiences. The sudden negative pressure changes that occur during the procedure, the stretching of the tissues, and the separation of the tube from the pleural tissue cause pain. This leads not only to physical discomfort but also to increased anxiety. Effectively controlling pain after surgical procedures is crucial for reducing complications and improving patient satisfaction. While pharmacological methods are often the first choice, interest in non-pharmacological approaches is increasing due to side effects and cost. In this context, rapid relaxation exercises and cold application are among the methods that are easy to implement, have no side effects, and have proven effective in nursing care. Rapid relaxation exercises are a simple breathing and muscle control technique that allows individuals to relax quickly by reducing muscle tension. This method balances the autonomic nervous system, producing both physiological and psychological relief. This helps reduce pain perception, control anxiety, and improve patient confidence. Cold application, on the other hand, reduces nerve conduction velocity by causing regional vasoconstriction and raises the pain threshold, providing an analgesic effect. Literature indicates that cold application is effective in reducing pain during invasive procedures such as chest tube removal and also increases patient satisfaction. Based on this information, the combined use of rapid relaxation exercise and cold application before chest tube removal may have a synergistic effect in reducing pain and anxiety. Furthermore, the noninvasiveness, ease of application, and cost-effectiveness of these methods provide significant advantages for nursing practice.This study was designed to determine the effects of rapid relaxation exercise and cold application before hest tube removal on pain, anxiety, and patient satisfaction.

DETAILED DESCRIPTION:
Open-heart surgery is a major surgical procedure frequently used in the treatment of cardiovascular diseases. After such operations, a chest tube is usually placed to drain air, fluid, and blood accumulated in the chest cavity. While a chest tube is vital in the postoperative period, it can cause intense pain, anxiety, and discomfort in patients during its removal. The literature reports that negative experiences during this process can significantly impact patient satisfaction, comfort, and overall well-being. The pain felt during chest tube removal is usually sudden, sharp, and short-lived; however, this pain can deepen the physical and psychological dimensions of the trauma experienced by the individual. Furthermore, increased anxiety can lead to undesirable physiological changes in cardiac patients, impairing hemodynamic stability. Therefore, investigating the effectiveness of non-invasive, low-cost, and easy-to-implement nursing interventions is crucial for improving the quality of patient care. Cold application (cryotherapy) and relaxation exercises are among the frequently used complementary methods to reduce pain and anxiety in the postoperative period. Cold application provides an analgesic effect by slowing nerve conduction; Rapid relaxation exercises, on the other hand, activate the parasympathetic nervous system, providing psychological relief. However, there is insufficient scientific evidence regarding the effectiveness of this technique during chest tube removal. Furthermore, randomized controlled trials examining the combined use of these interventions are limited. This study aimed to evaluate the effects of rapid relaxation exercises and cold application on pain, anxiety, and patient satisfaction before chest tube removal.

ELIGIBILITY:
Inclusion Criteria:

* Conscious, oriented, and cooperative.
* Can speak and understand Turkish.
* Does not have any psychiatric illness.
* Has a chest tube and is in a stable general condition.
* Has undergone a chest tube procedure for the first time.
* Is 18 years of age or older.
* Has not taken analgesics or sedatives 4 hours before the procedure.
* Has no vision or hearing problems.
* Volunteers to participate in the study.

Exclusion Criteria:

* Patients with any cognitive or psychological disorders
* Those who have had a chest tube placed before,
* Those who are on a mechanical ventilator (intubated),
* Those with chronic pain and routine painkiller use,
* Those with vision or hearing problems,
* Those who are taking analgesics immediately before chest tube removal.
* Patients who did not volunteer to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 15 minutes
  This scale, developed by Price et al. (1983), begins with 0 representing "no pain" and ends with 10 representing "unbearable pain." The patient is asked to score between 0 and 10 to express the severity of pain. The marked value represents the patient's pain score.
State Anxiety Inventory | 15 minutes
  This scale was developed by Spielberger et al. (1970) to measure the anxiety levels of individuals aged 14 and over. This study will use the 20-item "State Anxiety Inventory Scale" section of this two-section, 40-item scale. This Likert-type scale is rated according to the severity of the situation represented by the items: "not at all": 1, "a little": 2, "a lot": 3, and "completely": 4. This scale includes direct and reversed statements (items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20), and the scores for the reversed statements are calculated by converting them. Scores are adjusted so that 1 point = 4, 2 points = 3, 3 points = 2, and 4 points = 1. The scores for the other statements are taken as is and added. The anxiety score is obtained by subtracting the total score obtained from the reversed statements from the total score obtained for the direct statements and adding the predetermined constant value (the constant value for the state anxiety scale is 50). Possible scores for this i
Satisfaction Assessment Scale | 15 minutes
  This scale consists of a 10-cm vertical line without numbers to determine an individual's level of satisfaction. At one end of the line are the words "I am not satisfied at all" and at the other end are the words "I am very satisfied." The individual determines their level of satisfaction by considering all the components affecting them regarding the medical care provided and marks the point on the line corresponding to this state. The literature supports the use of this scale to measure satisfaction levels and has been reported to yield more reliable results. This scale will be used in the study to determine the level of satisfaction experienced by the individual with the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Unıversty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No